CLINICAL TRIAL: NCT02843685
Title: Regression Discontinuity Designs to Evaluate Real-world Effectiveness: a Case Study of Drotrecogin Alpha
Brief Title: Regression Discontinuity Design to Evaluate of Drotrecogin Alpha Effectiveness
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Allan J. Walkey, Assistant Professor of Medicine, Boston Medical Center
Other Study IDs: H-35010
Record Dates: First submitted 2016-07-15; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — drotrecogin alfa activated

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Drotrecogin alfa activated
  Other Names: Xigris

SUMMARY:
Many health care interventions and medications found to have benefits ("efficacy") in experimental, tightly-controlled, human research trials are later found to lack real-world health benefits ("effectiveness"). Inadequate surveillance of real-world clinical effectiveness may falsely reassure clinicians and those who monitor healthcare quality, propagating unrecognized ineffective or harmful treatments at high costs to patients and society. The failure to translate potential health benefits into realized gains, or to detect unexpected harms in healthcare delivery, stems from a lack of methods with which to robustly measure real-world (in)effectiveness. Current methods to detect changes in outcomes 'before and after' implementation may be biased by secular trends in healthcare practice and outcomes; other methods to compare outcomes for treated and untreated patients may be biased by unmeasured factors.

The current project aims to develop and demonstrate - as a proof-of-concept - the use of a quasi-experimental research method called 'regression discontinuity design (RDD)' in surveillance of real-world clinical effectiveness. RDD had previously found use in the evaluation of educational programs in which students scoring below a threshold were assigned an intervention. The US Department of Education considers RDD designs to have quality similar to randomized trials.

DETAILED DESCRIPTION:
Many health care interventions and medications found to have benefits ("efficacy") in experimental, tightly-controlled, human research trials are later found to lack real-world health benefits ("effectiveness"). Inadequate surveillance of real-world clinical effectiveness may falsely reassure clinicians and those who monitor healthcare quality, propagating unrecognized ineffective or harmful treatments at high costs to patients and society. The failure to translate potential health benefits into realized gains, or to detect unexpected harms in healthcare delivery, stems from a lack of methods with which to robustly measure real-world (in)effectiveness. Current methods to detect changes in outcomes 'before and after' implementation may be biased by secular trends in healthcare practice and outcomes; other methods to compare outcomes for treated and untreated patients may be biased by unmeasured factors.

The current project aims to develop and demonstrate - as a proof-of-concept - the use of a quasi-experimental research method called 'regression discontinuity design (RDD)' in surveillance of real-world clinical effectiveness. RDD had previously found use in the evaluation of educational programs in which students scoring below a threshold were assigned an intervention. The US Department of Education considers RDD designs to have quality similar to randomized trials. However, RDD has not been rigorously evaluated in the context of evaluating clinical effectiveness. RDD can be used whenever an intervention is given to patients scoring above a threshold on a continuous biomarker or risk score. This scenario often arises in clinical practice, in which thresholds are used to identify and treat 'high risk' patients. In RDD, outcomes are compared for patients just above and just below the threshold, who are similar, but receive different treatments.

The project will study the use of RDD in evaluating the real-world effectiveness of drotrecogin alpha, a medication that was recommended by the FDA to be given to critically ill patients with severe sepsis at high risk for mortality (APACHE score > 25). Drotrecogin alpha was shown to potentially have "effectiveness" using traditional methods of real-world research, but was eventually shown to not be clinically efficacious in subsequent large randomized trials. The present proposal is a 'proof-of-concept' study that will allow evaluation of effect estimates derived from RDD methods to those of gold standard, pooled randomized trial results. The demonstration of feasibility for a new research method, such as RDD, to evaluate real-world clinical effectiveness would be a major leap forward in the ability monitor for potential real world benefits and harms of new treatments.

ELIGIBILITY:
Inclusion Criteria:

* Included in PROGRESS severe sepsis registry

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An International Observational Study Among Severe Sepsis Patients Treated in the Intensive Care Unit (PROGRESS severe sepsis registry).
  The PROGRESS registry of severe sepsis cases is a unique resource that contains data linking APACHE scores, drotrecogin alpha administration, and hospital mortality outcomes, providing an opportunity to study RDD as a novel method of comparative effectiveness research, and compare results derived from RDD to prior studies using more traditional comparative effectiveness designs (i.e., propensity score adjustment).
Sampling Method: Non-Probability Sample
Enrollment: 12492 (Actual)
Dates: Start 2002-12; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Relative risk reduction for mortality | Duration of hospitalization, on average approximately 14 days
  The study will evaluate the change in the relationship between APACHE II scores and hospital mortality rate at the APACHE II threshold score of 25

SECONDARY OUTCOMES:
APACHE II scores at which drotrecogin alpha was used | Baseline
  Evaluation of drotrecogin alpha practice patterns at APACHE II score of 25
Change in mortality risk over time | 3 years
  The study will assess interaction between year and relative risk for mortality associated with drotrecogin alpha

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) is only available through consultation with the original PROGRESS registry study sponsor through https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Background] Martin G, Brunkhorst FM, Janes JM, Reinhart K, Sundin DP, Garnett K, Beale R. The international PROGRESS registry of patients with severe sepsis: drotrecogin alfa (activated) use and patient outcomes. Crit Care. 2009;13(3):R103. doi: 10.1186/cc7936. Epub 2009 Jun 30. PMID 19566927
- [Background] Beale R, Reinhart K, Brunkhorst FM, Dobb G, Levy M, Martin G, Martin C, Ramsey G, Silva E, Vallet B, Vincent JL, Janes JM, Sarwat S, Williams MD; PROGRESS Advisory Board. Promoting Global Research Excellence in Severe Sepsis (PROGRESS): lessons from an international sepsis registry. Infection. 2009 Jun;37(3):222-32. doi: 10.1007/s15010-008-8203-z. Epub 2009 Apr 28. PMID 19404580
- [Background] Walkey AJ, Bor J. Risk-based Heterogeneity of Treatment Effect in Trials and Implications for Surveillance of Clinical Effectiveness Using Regression Discontinuity Designs. Am J Respir Crit Care Med. 2015 Dec 1;192(11):1399. doi: 10.1164/rccm.201508-1533LE. No abstract available. PMID 26623693